CLINICAL TRIAL: NCT04265456
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Intravenous Pregabalin and Acetaminophen (Ofirmev®) in Healthy Volunteers
Brief Title: A Phase 1 Study to Evaluate Pregabalin and Acetaminophen in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nevakar, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CP-NVK009-0004
Record Dates: First submitted 2020-01-29; First posted 2020-02-11 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin; Prostaglandins B; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Up to 60 healthy male and female volunteers will be enrolled into one (1) of up to six (6) cohorts (n=10 per cohort).
  Within each cohort, subjects will be randomized at a ratio of 4:1 to receive IP (1300 mg of IV APAP plus a cohort specific dose of IV PGB) or placebo (saline) (8 active:2 placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1300 mg Acetaminophen and 100 mg IV Pregabalin (Experimental): The dose for the first cohort will be 1300 mg APAP and 100 mg PGB. For subsequent cohorts, the dose of APAP will remain constant at 1300 mg while the dose of PGB will be varied (will start with 100 mg TID and then based on tolerability will be either increased or decreased by 25 mg based on Safety Monitoring Committee decision).
  Interventions: Drug: Pregabalin 100mg; Drug: Acetaminophen 1300mg
- Placebo (No Intervention): Saline solution
- 1300 mg Acetaminophen and 100 mg +/- 25 IV Pregabalin (Experimental): Decisions to escalate or decrease the dose for Cohorts 2 through 6 will be dependent upon blinded review of emerging safety and tolerability data by the Safety Monitoring Committee (SMC). However, PK data is not part of the SMC review, but may be reviewed by a SMC designee at a later time.
  Interventions: Drug: Pregabalin 100mg; Drug: Acetaminophen 1300mg

INTERVENTIONS:
Drug: Pregabalin 100mg — Pregabalin is a structural derivative of the inhibitory neurotransmitter gamma aminobutyric acid with anticonvulsant, anxiolytic and sleep-modulating properties.
  Other Names: PGB
  Arms: 1300 mg Acetaminophen and 100 mg +/- 25 IV Pregabalin; 1300 mg Acetaminophen and 100 mg IV Pregabalin
Drug: Acetaminophen 1300mg — Acetaminophen is a non-salicylate antipyretic and non-opioid analgesic agent.
  Other Names: Ofirmev
  Arms: 1300 mg Acetaminophen and 100 mg +/- 25 IV Pregabalin; 1300 mg Acetaminophen and 100 mg IV Pregabalin

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single and multiple ascending dose study to determine a maximum tolerated dose of IV PGB and to evaluate the safety, tolerability, and PK of an admixture of IV PGB and a fixed dose of 1300 mg IV APAP in healthy adult volunteers.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, single and multiple ascending dose study to determine a maximum tolerated dose (MTD) of IV PGB and to evaluate the safety, tolerability, and PK of an admixture of IV PGB and a fixed dose of 1300 mg IV APAP in healthy adult volunteers.

Up to 60 subjects will be enrolled into one (1) of six (6) sequential cohorts (n=10 per cohort [8 APAP + PGB and 2 placebo]).

The dose for the first cohort will be 1300 mg APAP and 100 mg PGB. For subsequent cohorts, the dose of APAP will remain constant at 1300 mg while the dose of PGB will be varied (will start with 100 mg TID and then based on tolerability will be either increased or decreased by 25 mg) based on Safety Monitoring Committee decision.

The placebo will be the saline solution.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 55 years, inclusive at time of Screening
* Body mass index (BMI) between 18.5 and 28.0 kg/m2 inclusive, with a minimum weight of 50 kg and a maximum of 100 kg
* Healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination, and 12-lead ECG confirming normal sinus rhythm
* Negative tests for Hepatitis B surface antigen (HbsAg), hepatitis C virus antibody (anti-HCV), human immunodeficiency virus (HIV)-1 and HIV-2 antibody at Screening
* Routine clinical laboratory tests should be within normal limits at Screening and Admission (Day -1) or abnormalities deemed not clinically significant by the Investigator; for liver function tests, AST and ALT values should not be greater than 1.5 times the upper limit of normal range
* Negative screen for drugs of abuse or exhibit detectable alcohol levels by breathalyzer at the time of Screening or Admission
* Non-smokers or ex-smokers (must have ceased smoking ≥3 months prior Screening visit)

Female subjects:

* Must be of non-childbearing potential by surgical sterilization or postmenopausal OR Must not be pregnant, breast feeding, or planning to become pregnant AND must be practicing both a highly effective method of birth control from Screening until at least 90 days after the last dose of study drug.
* Women of childbearing potential must have a negative pregnancy test result at Screening and upon admission to the Clinical Trial Unit.

Exclusion Criteria:

* Has a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders
* Has a history of severe drug allergy, or severe hypersensitivity or severe food allergy, including anaphylaxis or known allergy or sensitivity to any component of PGB or APAP
* Has a history of alcoholism or drug abuse
* Has acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhea) at the time of Screening or Admission
* Consumption of drugs with enzyme-inducing properties, within 3 weeks prior to the initial dose of study drug and throughout the treatment phase
* Has used any prescription medicines, over the counter medicines, or herbal supplements, within 7 days of dosing
* Has used any investigational product or participated in any clinical trial within 30 days prior to Screening
* Has donated or received any blood or blood products within the 3 months prior to Screening;
* Not able to comply with the requirements of this study, including assessments, duration of admission of the study and expected follow up visits
* Is unwilling or unable to give written informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-07-22 (Actual)

PRIMARY OUTCOMES:
Treatment Related Adverse Events | 7 days
  The incidence and severity of treatment-emergent adverse events
Treatment related Drowsiness and Dizziness | 7 days
  The incidence and severity of somnolence and dizziness

SECONDARY OUTCOMES:
Plasma PK endpoints for APAP and PGB, SAD Phase, Cmax | 7 days
  Maximum observed concentration
Plasma PK endpoints for APAP and PGB, SAD Phase, Tmax | 7 days
  Time to maximum observed drug concentration (Tmax)
Plasma PK endpoints for APAP and PGB, SAD Phase, t1/2 | 7 days
  Apparent elimination half-life
Plasma PK endpoints for APAP and PGB, SAD Phase, AUC0-last | 7 days
  Area under the drug concentration-time curve from time zero to the last measurable concentration
Plasma PK endpoints for APAP and PGB, SAD Phase, AUC0-inf | 7 days
  AUC from time zero to infinity
Plasma PK endpoints for APAP and PGB, SAD Phase, λz | 7 days
  Apparent terminal elimination rate constant
Plasma PK endpoints for APAP and PGB, SAD Phase, CL | 7 days
  Apparent clearance
Plasma PK endpoints for APAP and PGB, SAD Phase, Vz | 7 days
  Apparent terminal volume of distribution
Plasma PK endpoints for APAP and PGB, multiple doses at steady state, AUCτ | 7 days
  Area under the plasma concentration-time curve during a dosage interval
Plasma PK endpoints for APAP and PGB, multiple doses at steady state, Tmax,ss | 7 days
  Time to Cmax at SS
Plasma PK endpoints for APAP and PGB, multiple doses at steady state, Cmax,ss | 7 days
  Maximum concentration at SS
Plasma PK endpoints for APAP and PGB, multiple doses at steady state, Cmin,ss | 7 dyas
  Minimum concentration at ss
Plasma PK endpoints for APAP and PGB, multiple doses at steady state, Cav,ss | 7 days
  Average plasma concentration at SS
Plasma PK endpoints for APAP and PGB, multiple doses at steady state, Vz, ss | 7 days
  Apparent volume of distribution at SS
Plasma PK endpoints for APAP and PGB, multiple doses at steady state, CLss | 7 days
  Apparent total clearance at SS
Plasma PK endpoints for APAP and PGB, multiple doses at steady state, λz,ss | 7 days
  Apparent first order terminal elimination rate constant at steady state
Plasma PK endpoints for APAP and PGB, multiple doses at steady state, R | 7 days
  Accumulation index
Plasma PK endpoints for APAP and PGB, multiple doses at steady state, LF | 7 days
  Linearity factor
Plasma PK endpoints for APAP and PGB, multiple doses at steady state | 7 days
  Fluctuation ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Lotus Clinical Resarch,LLC, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No